CLINICAL TRIAL: NCT05689398
Title: Rehabilitation on Equal Terms - A Study Focusing on Recovery and Mortality of Migrated Women With Breast Cancer: The ReMig Study
Brief Title: Rehabilitation on Equal Terms - The ReMig Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: ReMig
Record Dates: First submitted 2022-11-29; First posted 2023-01-19 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: Rehabilitation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The ReMig-study aims to increase knowledge about rehabilitation needs, the rehabilitation process of arabic-speaking migrated women with BC, to increase the prerequisites for optimized and equal cancer care. The study aims to map migrated Arabic-speaking women's breast cancer rehabilitation with a focus on mental and physical recovery, lifestyle habits as well as satisfaction and goals with the rehabilitation and compare these outcomes with the outcomes of Swedish-speaking women. Further aim is to explore migrated Arabic-speaking women´s experiences and attitudes towards breast cancer rehabilitation.

DETAILED DESCRIPTION:
Annually, over 2 million women are diagnosed with breast cancer (BC) globally, of which about 8300 in Sweden. Today, 20% of the Swedish population is foreign born and previous research has shown that women who have migrated are particularly vulnerable when diagnosed with BC. Research focusing on migrated women is sparse as they are often excluded from research, but available research shows that experience and management of BC differs depending on ethnicity, that the women to a lesser extent participate in BC screening and rehabilitation and that they have a higher mortality than Swedish born women. In recent years, measures to promote early BC diagnosis have been initiated, but knowledge of how optimized rehabilitation should be ensured to promote recovery and reduce the socioeconomic burden is lacking.

This study aims to map the rehabilitation of migrant Arabic-speaking women with a focus on mental and physical recovery, lifestyle habits and satisfaction and goals with the rehabilitation in the first year after BC diagnosis and compare these outcomes with Swedish-speaking women. Further to elucidate migrated Arabic-speaking women´s experiences and attitudes towards breast cancer rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Undergone treatment for primary breast cancer
* ≤18 years old
* Ability to communicate in the Arabic language
* Written informed consent

Exclusion Criteria:

* Recurrent disease
* Palliative diagnosis
* Pregnancy
* Prior history of breast cancer
* Inability to participate in the study due to cognitive impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are planned to be recruited at breast cancer clinics in southern Sweden. The selection is coming to consist of Arabic-speaking women, ≤18 years of age who have migrated to Sweden and who have been diagnosed with BC (N=140). To this data comes a matched sample with data for Swedish-speaking women from the ReScreen study (dnr 201/505) to be used as a basis for the comparative analyses.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Psychological Distress | 1 week pre-operative, after surgery at 2 weeks, 3 ,6 ,9 and 12 months postoperative. Evaluating change over time.
  Psychological Distress measured by the "Distress thermometer". A instrument that the patients answer themselves measuring the level of distress and the potential problems the may have.
General Quality of life | 1 week pre-operative, after surgery at 2 weeks, 3 ,6 ,9 and 12 months postoperative. Evaluating change over time.
  The instrument EORTC Core Quality of Life questionnaire (QLQ-C30), developed by the EORTC (European Organization for Research and Treatment of Cancer) and measures quality of life. The QLQ-C30 is composed of both multi-item scales and single-item measures (total 28 questions)
  , including. five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures transforms to range in score from 0 to 100. A high scale score represents a higher response level, which means that a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Breast cancer specific quality of life | 1 week pre-operative, after surgery at 2 weeks, 3 ,6 ,9 and 12 months postoperative. Evaluating change over time.
  The instrument QLQ-BR23 is developed by the EORTC (European Organization for Research and Treatment of Cancer) and measures diagnose specific quality of life. The QLQ-BR23 includes five multi-item scales to assess body image, sexual functioning, systemic therapy side effects, breast symptoms, and arm symptoms. Additionally, single items assess sexual enjoyment, future perspective and being upset by hair loss. The range in score from 0 to 100. A high score for the functional scales represents a high/healthy level of functioning, while a high score for the symptom scales represents a high level of symptomatology or problems.
Resilience | 1 week pre-operative, after surgery at 2 weeks, 3 ,6 ,9 and 12 months postoperative. Evaluating change over time.
  Connor-Davidson Resilience scale (CD-RISC) will be used to measure patients resilience trough 25 questions ranging from 0-4. Lower scores indicates more problems. Scoring of the scale CD-RISC-25 is based on summing the total of all items, each of which is scored from 0-4, the full range is from 0 to 100, with higher scores reflecting greater resilience.
Body mass index | 1 week pre-operative, 6 ,9 and 12 months postoperative. Evaluating change over time.
  Body mass index, based on weight (in kilograms) and height (in meters). Weight and height will be combined to report BMI in kg/m^2. Height will be reported only at baseline (eg. 1 week pre-operative) and weight at baseline (1 week pre-operative), 6 ,9 and 12 months postoperative.
Working status/sick leave | 1 week pre-operative,after surgery at 2 weeks, 3 ,6 ,9 and 12 months postoperative. Evaluating change over time.
  Sick leave may indicate that the woman experience more complications of the surgery or /and cancer treatment. Follow-up question regarding the extent in percent of the sickleave.
Physical activity/life style | 1 week pre-operative,after surgery at 2 weeks, 3 ,6 ,9 and 12 months postoperative. Evaluating change over time.
  Four questions regarding life style and physical activity. The questions is about the amount of time per week the woman is performing physical activity with high intensity, performing physical activity with low intensity, the grade of physical strenuous of work or daily activities and the hours spent sedentary. The answer options is given in minutes from 0 up to more than 300 minutes for physical activity respectively from 0 minutes to more than 8 hours for time spent sedentary.
Rehabilitation process | After surgery at 6 ,9 and 12 months postoperative. Evaluating change over time.
  Questions regarding the experiences of the rehabilitation process, the extent of information, the extent of participation in decisions regarding rehabilitation,support from healthcare and the satisfaction of recovery and rehabilitation. The answer options range from not at all to a very high extent.

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University, Skåne university hospital, Helsingborgs sjukhus, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No